CLINICAL TRIAL: NCT02233205
Title: Safety Study of Combining Ultrasound Microbubbles and Chemotherapy to Treat Malignant Neoplasms of Liver Metastases From Gastrointestinal Tumors and Pancreatic Carcinoma
Brief Title: Safety Study of Combining Ultrasound Microbubbles and Chemotherapy to Treat Malignant Neoplasms of Digestive System
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Kun Yan, chief director, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014YJZ11
Record Dates: First submitted 2014-08-31; First posted 2014-09-08 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Gastrointestinal Neoplasms
Keywords: microbubble; chemotherapy; alimentary
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Platinum; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- microbubbles & platinum and gemcitabine (Experimental): In 30min after chemotherapy, inject ultrasonic microbubbles 1 ml once and inject 5 times in 20min and locate the ultrasonic probe on the lesion The chemotherapy of pancreatic is gemcitabine.The chemotherapy of liver metastases is oxaliplatin with taxol.
  Interventions: Device: ultrasonic microbubbles; Drug: platinum and gemcitabine

INTERVENTIONS:
Device: ultrasonic microbubbles — inject 1ml once and five times in 20min, locate the probe on the lesion at the same time
  Other Names: Sonovue
Drug: platinum and gemcitabine — Chemotherapy drug of pancreatic carcinoma is gemcitabine. Chemotherapy drug of liver metastases is oxaliplatin and taxol.

SUMMARY:
Ultrasonic sonoporation can increase the release of chemotherapeutics, thus increasing the therapeutic effects. The main purpose is to identify the safety of combining ultrasonic microbubbles and chemotherapeutics to treat malignant neoplasms of hepatic metastases from alimentary system and pancreatic carcinoma.

DETAILED DESCRIPTION:
Ultrasonic sonoporation can increase the release of chemotherapeutics, thus increasing the therapeutic effects.

1. Main purpose

   1. To identify the safety of combining ultrasonic microbubbles and chemotherapeutics to treat malignant neoplasms of hepatic metastases from alimentary system and pancreatic carcinoma.
   2. To explore the largest mechanical index and ultrasonic treatment time which patients can endure.
2. Secondary purpose

   1. To observe tumor clinical benefit rate (CR+PR+SD).
   2. To evaluate the preliminary effect,such as time to failure(TTF), time to death(TTD)

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of liver metastases from alimentary system and pancreatic carcinoma
* Failed routine chemotherapy
* Neoplasms can be evaluated by imaging
* ECOG《2

Exclusion Criteria:

* Have systematic chemotherapy in 2 weeks
* Be allergic to ultrasonic microbubbles and chemotherapeutics
* Uncontrolled high blood pressure, cardiovascular disease
* Active bleeding
* Have serious mental and psychological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 1 month

SECONDARY OUTCOMES:
Time to Disease Progression | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kun Yan, Master, Principal Investigator — Peking University Cancer Hospital & Institute; Lin Shen, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

REFERENCES:
- [Result] Kotopoulis S, Dimcevski G, Gilja OH, Hoem D, Postema M. Treatment of human pancreatic cancer using combined ultrasound, microbubbles, and gemcitabine: a clinical case study. Med Phys. 2013 Jul;40(7):072902. doi: 10.1118/1.4808149. PMID 23822453
- [Result] Dewitte H, Van Lint S, Heirman C, Thielemans K, De Smedt SC, Breckpot K, Lentacker I. The potential of antigen and TriMix sonoporation using mRNA-loaded microbubbles for ultrasound-triggered cancer immunotherapy. J Control Release. 2014 Nov 28;194:28-36. doi: 10.1016/j.jconrel.2014.08.011. Epub 2014 Aug 22. PMID 25151979
- [Result] Fan Z, Kumon RE, Deng CX. Mechanisms of microbubble-facilitated sonoporation for drug and gene delivery. Ther Deliv. 2014 Apr;5(4):467-86. doi: 10.4155/tde.14.10. No abstract available. PMID 24856171
- [Result] Feichtinger GA, Hofmann AT, Slezak P, Schuetzenberger S, Kaipel M, Schwartz E, Neef A, Nomikou N, Nau T, van Griensven M, McHale AP, Redl H. Sonoporation increases therapeutic efficacy of inducible and constitutive BMP2/7 in vivo gene delivery. Hum Gene Ther Methods. 2014 Feb;25(1):57-71. doi: 10.1089/hgtb.2013.113. Epub 2013 Nov 27. PMID 24164605